CLINICAL TRIAL: NCT01158001
Title: Telemedicine for Improved Delivery of Psychosocial Treatments for Post Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 080513; PT074431
Record Dates: First submitted 2009-02-20; First posted 2010-07-08 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Posttraumatic Stress Disorders; Depression; Anxiety
Keywords: Posttraumatic stress disorders; Telemedicine; Psychotherapy; Neuropsychological test; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychotherapy via telemedicine (Experimental): In this arm, veterans received standard psychotherapy (prolonged exposure therapy) in a novel format - interacting with a therapist via videoconferencing.
  Interventions: Behavioral: Prolonged exposure therapy
- Face-to-face (in person) psychotherapy (Active Comparator): In this arm, veterans received standard psychotherapy (prolonged exposure therapy) in the traditional format - in person with a therapist.
  Interventions: Behavioral: Prolonged exposure therapy

INTERVENTIONS:
Behavioral: Prolonged exposure therapy — Twelve sessions (90 minutes each) of prolonged exposure therapy

SUMMARY:
The objective of the proposed study is to conduct a systematic comparison of post traumatic stress disorder (PTSD) outcomes for veterans receiving exposure therapy via telemedicine versus in-person care. The primary aim is to determine feasibility: whether telemedicine can be used as a tool to extend effective, specialized mental health services, such as Prolonged Exposure therapy (PE; a therapy designed to help clients face fears related to a traumatic event), to veterans with limited access to care. A secondary aim is to determine if therapy delivered by telemedicine affects the quality of care in terms of clinical outcomes and the quality of patient-therapist interaction. A tertiary aim is to examine whether results from neuropsychological testing predict treatment outcomes.

DETAILED DESCRIPTION:
The objective of the proposed study is to conduct a systematic comparison of post traumatic stress disorder (PTSD) outcomes for veterans receiving exposure therapy via telemedicine versus in-person care. Specifically, prolonged exposure therapy (PE) was conducted with veterans individually, either in person or via videoconferencing technology. PE is designed to help clients face fears related to a traumatic experience by guiding individuals through exposures to the memory of the event (called "imaginal exposure") and exposures to feared situations (called "in vivo" exposures).

The primary aim is to determine the feasibility of whether telemedicine can be used as a tool to extend effective, specialized mental health services, such as PE to veterans with limited access to care. This is measured in part through patient and therapist satisfaction ratings in each condition.

A secondary aim is to determine if therapy delivered by telemedicine affects the quality of care in terms of clinical outcomes and the quality of patient-therapist interaction. This is measured by relative changes in symptoms, primarily in PTSD, depressive symptoms, and anxiety symptoms.

A tertiary aim is to examine whether results from neuropsychological testing predict treatment outcomes across conditions. This includes seven measures of executive functioning. The hypothesis is that poorer performance on these measures may be associated with less improvement on measures of symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of chronic PTSD due to combat; comorbid mood and anxiety disorders are expected, and will be permitted (to maximize generalizability) if PTSD symptoms are judged to be predominant based on primacy and severity of symptoms
* Age 18 or older
* English literacy

Exclusion Criteria:

* Unmanaged psychosis or manic episodes in past year
* Concurrent psychotherapies targeting PTSD or depression or that entail exposure therapy [veterans who are engaged in treatment for non-PTSD symptoms (e.g., 12-step programs for substance problems) will be eligible]
* Severe cardiovascular or respiratory disease that would make it difficult to ensure regular attendance at psychotherapy sessions
* Probable dementia; OR
* Head trauma resulting in loss of consciousness longer than 20 minutes. Potential participants who have had changes in the type and dosage of psychotropic medications in the preceding two months will be asked to wait until their medication regimen has stabilized to minimize treatment confounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Clinician-administered PTSD Scale (CAPS) diagnostic interview | Pre-treatment, post-treatment (14 weeks after pre-treatment assessment), follow-up six months after post-treatment assessment
  Measure of PTSD diagnosis and severity

SECONDARY OUTCOMES:
PHQ-9 (self-reported depression) | Pre-treatment, weekly during 12 weeks of treatment, post-treatment (14 weeks after pre-treatment assessment), follow-up six months after post-treatment assessment
  Measure of depressive symptoms
PTSD Checklist (PCL; self-reported PTSD symptoms) | Pre-treatment, weekly during 12 weeks of treatment, post-treatment (14 weeks after pre-treatment assessment), follow-up six months after post-treatment assessment
  Measure of 17 posttraumatic stress disorder (PTSD) symptoms from specific event (PCL-S)
Neuropsychological testing battery to assess cognitive functioning | Pre-treatment and post-treatment (14 weeks after pre-treatment assessment)
  1. Wechsler Test of Adult Reading
  2. Rey Complex Figure task
  3. California Verbal Learning Test
  4. Wisconsin Card Sort Test
  5. Wechsler Adult Intelligence Scale Digit Span
  6. Delis-Kaplan Executive Functioning System (D-KEFS) Verbal Fluency
  7. Delis-Kaplan Executive Functioning System (D-KEFS) Color-Word Interference
  8. Delis-Kaplan Executive Functioning System (D-KEFS) Trails

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Thorp, PhD, Principal Investigator — Veterans Affairs San Diego Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States